CLINICAL TRIAL: NCT00396019
Title: A Phase II Trial of Peginterferon Alfa-2b (PEG-Intron) for Plexiform Neurofibromas
Brief Title: Study of PEG-Intron for Plexiform Neurofibromas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jean M. Tersak, M.D., Associate Professor of Pediatrics, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 06-116; NCT00678951 (obsolete NCT alias)
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Plexiform Neurofibroma
MeSH Terms: conditions — Neurofibroma, Plexiform | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PEG-Intron

SUMMARY:
This study is for slow growing tumors called plexiform neurofibromas (PNF) which are a relatively common problem in people with neurofibromatosis type 1 (NF1). These tumors are benign but as they grow, they can become disfiguring as well as disabling or even life threatening. They often cause pain, difficulty using arms or legs because of spinal cord compression, and/or nerve damage. At present, the only available therapy for plexiform neurofibromas is to try to surgically remove as much of the tumor as is possible. Because these tumors grow into the surrounding areas, total surgical resection is often impossible. Most tumors will re-grow after surgery if the entire tumor cannot be removed. To date, other treatments including chemotherapy and radiotherapy have not been able to shrink these tumors.

Interferon is a drug that is used for different types of tumors as well as for hepatitis. It has been used in the treatment of plexiform neurofibromas (PNF) with some subjects showing improvement in symptoms and/or a decrease in the size of the tumor. Most subjects had no further growth of their tumor while on the PEG-Intron. The drug used in this study is PEG (pegylated)-Intron. PEG-Intron is a long acting form of interferon which keeps the drug from being broken down in the body for a longer period of time and potentially could be more effective than the short-acting interferon. PEG-Intron has been approved by the Food and Drug Administration (FDA) for the treatment of Hepatitis C.

The goals of this study are:

1. To determine how your child's plexiform neurofibroma responds to PEG-Intron when given weekly.
2. To determine the side effects of PEG-Intron when given weekly to participants with plexiform neurofibromas.
3. To evaluate a new method of measuring changes in the size of tumors called volume analysis. This method measures the entire volume of a tumor in three dimensions. The standard method of measuring tumors uses only the length and/or width of the tumor. By studying the different ways of measuring tumors the investigators hope to be able to determine which method is the most accurate and useful.

DETAILED DESCRIPTION:
PEG-Intron will be given every week through a small needle under the skin, in the same way that insulin is given to people with diabetes. Subjects will be taught to do this at home. As long as the tumor isn't growing and the side effects are tolerable, the injections will be given once a week for 2 years.

Children will be enrolled on the study into one of three strata (patient groups): strata 1 includes children who do not have any symptoms associated with their PNF and MRI scans over the past year may or may not show tumor growth, strata 2 includes children who have symptoms associated with the PNF but MRI scans over the past year have not shown growth and strata 3 includes children who have shown an increase in the size of the PNF on MRI scans over the past year, with or without any symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 months to 21 years
* Diagnosis Patients with NF1 and progressive, symptomatic or life-threatening plexiform neurofibromas which are not surgically resectable. Patients without biopsy-proof of plexiform must have at least one other diagnostic criteria for NF1: 6 or more cafe-au-lait spots, freckling in the axilla or groin, optic glioma, 2 or more Lisch nodules, distinctive bony lesion, first degree relative with NF1.
* Only eligible if complete tumor resection is not feasible, or if a patient with a surgical option refuses surgery.
* Patients may be treated on this trial without having received prior therapy. If patients have received prior therapy, they must have recovered from all toxic effects prior to entering this study.
* Must have life expectancy of at least 12 months and a performance score (Karnofsky or Lansky) of > or equal to 50.
* Must have adequate liver, kidney and bone marrow function

Exclusion Criteria:

* Clinically significant unrelated systemic illness.
* Received an investigational agent within the past 30 days.
* Evidence of active visual pathway glioma
* History of malignant peripheral nerve sheath tumor or ther cancer other than surgically cured non-melanoma skin cancer or cervical carcinoma in situ
* Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumor, or immunotherapy.
* Inability to return for follow-up visits or obtain follow-up studies
* Severe cardiovascular disease
* Pre-existing sever psychiatric condition or history of psychiatric disorder requiring hospitalization or a history of suicidal ideation or attempt.
* Thyroid dysfunction not responsive to therapy.
* Uncontrolled diabetes mellitus
* History of seropositivity for HIV
* Subjects who are pregnant, lactating, or of reproductive potential and not practicing an effective means of contraception.
* Any medical condition requiring chronic systemic corticosteroids.
* Subjects who are known to be actively abusing alcohol or drugs.

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tersak, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Jakacki RI, Dombi E, Steinberg SM, Goldman S, Kieran MW, Ullrich NJ, Pollack IF, Goodwin A, Manley PE, Fangusaro J, Allen R, Widemann BC. Phase II trial of pegylated interferon alfa-2b in young patients with neurofibromatosis type 1 and unresectable plexiform neurofibromas. Neuro Oncol. 2017 Feb 1;19(2):289-297. doi: 10.1093/neuonc/now158. PMID 27510726

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum 1 No Symptom With or Withour Tumor Growth; Stratum 2 Symptoms no Tumor Growth; Stratum 3 Tumor Growth With or Without Symptoms: Peg-intron given every week
Period: Overall Study
Arm/Group | Stratum 1 No Symptom With or Withour Tumor Growth | Stratum 2 Symptoms no Tumor Growth | Stratum 3 Tumor Growth With or Without Symptoms
Started | 27 | 29 | 30
Completed | 27 | 26 | 29
Not Completed | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 No Symptom With or Withour Tumor Growth | Stratum 2 Symptoms no Tumor Growth | Stratum 3 Tumor Growth With or Without Symptoms | Total
Number analyzed (Participants) | 27 | 26 | 29 | 82
Age, Customized [Count of Participants; unit: Participants] — Population: Age data is missing for one subject.
  Participants
    Less than 5 years: number analyzed (Participants) | 27 | 25 | 29 | 81
    Less than 5 years | 3 | 8 | 9 | 20
    5 to 12 years: number analyzed (Participants) | 27 | 25 | 29 | 81
    5 to 12 years | 10 | 9 | 12 | 31
    greater than or equal to 12 years: number analyzed (Participants) | 27 | 25 | 29 | 81
    greater than or equal to 12 years | 14 | 8 | 8 | 30
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data was not captured with demographic/enrollment data.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 29 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Imaging Response in Strata 1 and 2
Description: A response was defined as a ≥20% reduction in the sum of the volume of the "target" plexiform neurofibroma ( PN) within 12 months confirmed by a follow-up MRI after ≥4 weeks.
Time Frame: MRI scans were performed at baseline and at months 4, 8, 12, 18, and 24 while on treatment and every 6 months thereafter until off study.
Measure: Number; unit: participants
Arm/Group | Stratum 1 No Symptom With or Withour Tumor Growth | Stratum 2 Symptoms no Tumor Growth
Number analyzed (Participants) | 27 | 26
participants
  Confirmed Response | 0 | 1
  Unconfirmed Response | 1 | 0

2. Primary Outcome: Clinical Response in Stratum 2
Description: Clinical response was defined as a protocol-specified improvement in ophthalmologic evaluation, an improvement of at least one level in performance status (PS) ≥50% decrease in the amount of pain medications required per week compared with baseline or ability to change from a narcotic to a nonnarcotic analgesic, sustained for at least one month.
Time Frame: baseline, week 6, months 4, 8, 12, 18, and 24 while on treatment and every 6 months thereafter until off study
Population: Only participants in Stratum 2 contributed data for this Outcome Measure
Measure: Number; unit: participants
Groups:
- Stratum 2 Symptoms on Tumor Growth: Peg-intron given every week
Arm/Group | Stratum 2 Symptoms on Tumor Growth
Number analyzed (Participants) | 26
participants | 3

3. Primary Outcome: Time to Progression (TTP) in Stratum 3
Description: TTP was estimated by the Kaplan-Meter method
Time Frame: baseline, week 6, months 4, 8, 12, 18, and 24 while on treatment and every 6 months thereafter until off study
Population: Only participants in Stratum 3 contributed data for this Outcome Measure
Measure: Median (Full Range); unit: months
Groups:
- Stratum 3: Tumor Growth With or Without Symptoms: Peg-intron given every week
Arm/Group | Stratum 3: Tumor Growth With or Without Symptoms
Number analyzed (Participants) | 29
months | 29.4 [7.1 to NA] — ¹not everyone experienced endpoint

4. Secondary Outcome: Number of Participants With Imaging Response in Stratum 3
Description: A Response was defined as a ≥ 20% reduction in the sum of the volume of the "target" plexiform neurofibroma (PN) within 12 months, confirmed by a follow-up MRI after ≥ 24 weeks
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Stratum 3: Tumor Growth With or Without Symptoms
Number analyzed (Participants) | 29
participants
  Confirmed Response | 1
  Unconfirmed Response | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during clinic visits at baseline, week 6, months 4, 8, 12, 18, and 24 while on treatment and every 6 months thereafter until off study
Description: Other
Arm/Group | Stratum 1 No Symptom With or Withour Tumor Growth | Stratum 2 Symptoms no Tumor Growth | Stratum 3 Tumor Growth With or Without Symptoms
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 7/27 | 8/26 | 6/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 No Symptom With or Withour Tumor Growth (N=27) | Stratum 2 Symptoms no Tumor Growth (N=26) | Stratum 3 Tumor Growth With or Without Symptoms (N=29)
Fatigue (General disorders) | 2 | 4 | 2
Behavior (Psychiatric disorders) | 2 | 3 | 2 — Behavior
Allergic Reaction (General disorders) | 1 | 0 | 0 — Allergic Reaction
Depression (Psychiatric disorders) | 2 | 1 | 0 — Worsening depression
Transaminitis (Investigations) | 0 | 0 | 2 — Transaminitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No